CLINICAL TRIAL: NCT03247946
Title: The Influence of Upright Feeding Position on Pulmonary and Ear Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Avital Avraham, Principal investigator, Associate Professor, Institute of Pulmonology, email: avital@hadassah.org.il, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0349-10-HMO
Record Dates: First submitted 2017-08-03; First posted 2017-08-14 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Feeding and Eating Disorders
Keywords: infant; feeding position; respiratory; ear
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: 3 month old infants were recruited from 2 Mother-Child-Health clinics and followed for 12 months. Mothers from intervention group were instructed to feed their babies (88 infants) with their head in upright position. Mothers from control group (75 infants) fed their infant regularly without any instructions . Respiratory and ear morbidity were evaluated during the following 12 month period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): intervention: upright head position
  Interventions: Behavioral: upright head position
- Control group (No Intervention): no feeding position instructions

INTERVENTIONS:
Behavioral: upright head position — Bottle feeding of infants with their head in upward and not supine head position
  Arms: Intervention group

SUMMARY:
Does upright feeding position of 3 month old infants reduce respiratory and ear morbidity during the following year?

DETAILED DESCRIPTION:
The investigators examined the influence of teaching mothers to feed infants with their head in an upright position and evaluated the infant ear and respiratory morbidity during a one-year follow-up. Mothers of 88 infants born during 2011 were instructed by trained nurses at Maternal-Child-Health clinics to feed their infants with their head in upright position (intervention group). The control group consisted of 75 mothers of infants of similar socioeconomic background who fed their infant regularly without any instructions and were followed at another Maternal-Child-Health clinic. Feeding position was evaluated at the beginning and the end of the study, and morbidity data of both groups were evaluated at every 3-month follow-up meeting. The study was part of the PhD thesis of Efrat Danino, Head Nurse of Pediatric Department at Hadassah Medical Organization.

ELIGIBILITY:
Inclusion Criteria:

* healthy 3 month old infants, bottle fed at least once a day, parent agreeing to participate

Exclusion Criteria:

* Prematurity, need of supplemental oxygen, broncho-pulmonary dysplasia, cystic fibrosis, familial dysautonomia, cleft lip or cleft palate, any ear-throat-lung or airway congenital anomaly, congenital heart disease, any other chronic disease of childhood or malignancy

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2012-08-19 (Actual); Study Completion 2012-08-19 (Actual)

PRIMARY OUTCOMES:
Infant morbidity | every 12 weeks visit to Mother Child Health clinic until end of 1 year follow up
  respiratory (cough, wheezing, physician diagnosed bronchitis or pneumonia), ear (OM, SOM), prolonged fever, use of antibiotics and inhalations.

SECONDARY OUTCOMES:
Feeding position angle | at beginning and end of study (1 year follow up)
  description of feeding position angle

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tully SB, Bar-Haim Y, Bradley RL. Abnormal tympanography after supine bottle feeding. J Pediatr. 1995 Jun;126(6):S105-11. doi: 10.1016/s0022-3476(95)90249-x. PMID 7776069